CLINICAL TRIAL: NCT05731895
Title: Pharmacokinetics, Safety and Tolerability of BI 425809 (Iclepertin) Following Oral Administration in Male and Female Participants With Different Degrees of Hepatic Impairment (Child-Pugh Classification A and B) Compared With Matched Male and Female Participants With Normal Hepatic Function (an Open-label, Non-randomised, Single-dose, Parallel, Individualmatched Design Trial)
Brief Title: A Study to Test How Iclepertin is Taken up in the Blood of People With and Without Liver Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0048; 2022-003418-35 (EudraCT Number)
Record Dates: First submitted 2023-02-08; First posted 2023-02-16 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — BI 425809

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Participants with mild hepatic impairment (Child-Pugh A) (Experimental)
  Interventions: Drug: BI 425809 (iclepertin)
- Arm 2: Participants with moderate hepatic impairment (Child-Pugh B) (Experimental)
  Interventions: Drug: BI 425809 (iclepertin)
- Arm 3: Participants with normal hepatic function individually matched to participants of Arm 1 (Experimental)
  Interventions: Drug: BI 425809 (iclepertin)
- Arm 4: Participants with normal hepatic function individually matched to participants of Arm 2 (Experimental)
  Interventions: Drug: BI 425809 (iclepertin)

INTERVENTIONS:
Drug: BI 425809 (iclepertin) — BI 425809 (iclepertin)

SUMMARY:
This study is open to people with and without liver problems. People can join the study if they are 18 to 79 years of age and have a body mass index (BMI) between 18.5 and 35 kg/m2.

Iclepertin (also called BI 425809) is a medicine that is being developed to treat diseases of the brain. The purpose of this study is to find out whether having liver problems influences how iclepertin is taken up in the body. All participants take iclepertin once as a tablet.

Participants are in the study for 2 to 3 weeks. During the first part of the study, they stay at the study site for 4 nights. Afterwards, there are 5 visits to the study site and 1 call. The site staff measures the amount of iclepertin in the blood. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

Inclusion criteria applicable to all participants:

* Male or female participants
* Age 18-79 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 35 kilograms per meter squared (kg/m2) (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male participants are not required to use contraception
* Women of childbearing potential are allowed to participate provided they use a highly effective contraception from at least 30 days before the administration of trial medication until 30 days after trial completion.

The following methods of contraception are considered adequate for female participants of childbearing potential:

* Use of combined (oestrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
* Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
* Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
* Sexually abstinent (true abstinence, in line with the preferred and usual lifestyle of the subject) - -A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant.

Female participants are not considered to be of childbearing potential if they are either surgically sterilized (including hysterectomy) or postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle-stimulating hormone (FSH) above 40 unit per liter (U/L) and oestradiol below 30 nanogram per liter (ng/L) is confirmatory).

Inclusion criteria applying only to participants with impaired hepatic function:

* Hepatic impairment classified as Child-Pugh A (score 5-6 points) or Child Pugh B (score 7-9 points)
* further inclusion criteria apply

Inclusion criteria applying only to participants with normal hepatic function:

* Individually matched to participants with hepatic impairment according to sex, age, and weight
* further inclusion criteria apply

Exclusion criteria

Exclusion criteria applying to all participants:

* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* For diabetics only: uncontrolled diabetes mellitus with a glycated hemoglobin (HbA1c) > 9
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics (PK) of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the Central Nervous System (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder or history of suicide attempts)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections
* further exclusion criteria apply

Exclusion criteria applying only to participants with hepatic impairment:

* A marked prolongation of the time from the start of the Q wave to the end of the T wave (QT)/ Corrected QT (QTc) interval (such as QTc Fridericia (QTcF) intervals that are repeatedly greater than 480 milliseconds (ms) in males or repeatedly greater than 500 ms in females) or any other clinically relevant electrocardiogram (ECG) finding at screening
* further exclusion criteria apply

Exclusion criteria applying only to participants with normal hepatic function:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
* further exclusion criteria apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of iclepertin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 9 days
Maximum measured concentration of iclepertin in plasma (Cmax) | Up to 9 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of iclepertin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 9 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com